CLINICAL TRIAL: NCT02609646
Title: Antibiotic Pharmacokinetics in Critically Ill Patients
Brief Title: AbioKin - Antibiotic Kinetics
Status: Completed | Type: Observational
Sponsor: Gruppo Italiano per la Valutazione degli Interventi in Terapia Intensiva (Other)
Responsible Party: Sponsor
Other Study IDs: AbioKin
Record Dates: First submitted 2015-11-18; First posted 2015-11-20 (Estimated); Last update posted 2021-01-19 (Actual); Status verified 2016-07

CONDITIONS: Critical Illness; Infection
Keywords: Anti-Infective Agents; Pharmacokinetics; Critically ill patients
MeSH Terms: conditions — Critical Illness; Infections | interventions — Linezolid; Meropenem; Piperacillin, Tazobactam Drug Combination; Vancomycin

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples to measure antibiotic plasma concentration
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- linezolid: patients treated with linezolid
  Interventions: Drug: Linezolid
- meropenem: patients treated with meropenem
  Interventions: Drug: Meropenem
- piperacillin/tazobactam: patients treated with piperacillin/tazobactam
  Interventions: Drug: Piperacillin-tazobactam combination product
- vancomycin: patients treated with vancomycin
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Linezolid — Drug choice is performed according to standard clinical practice, that will not be modified by the participation in the study. As a consequence, assignment of patients to groups is not protocol based, but it is defined by standard clinical choices.
  Groups: linezolid
Drug: Meropenem — Drug choice is performed according to standard clinical practice, that will not be modified by the participation in the study. As a consequence, assignment of patients to groups is not protocol based, but it is defined by standard clinical choices.
  Groups: meropenem
Drug: Piperacillin-tazobactam combination product — Drug choice is performed according to standard clinical practice, that will not be modified by the participation in the study. As a consequence, assignment of patients to groups is not protocol based, but it is defined by standard clinical choices.
  Groups: piperacillin/tazobactam
Drug: Vancomycin — Drug choice is performed according to standard clinical practice, that will not be modified by the participation in the study. As a consequence, assignment of patients to groups is not protocol based, but it is defined by standard clinical choices.
  Groups: vancomycin

SUMMARY:
The purpose of this study is to investigate the pharmacokinetic properties in critically ill patients of a few of the most used antimicrobial drugs (amikacin, linezolid, meropenem, piperacillin/tazobactam, vancomycin). The primary objective is the identification of the clinical parameters affecting the kinetics of these drugs and the study of the contribution of extracorporeal depuration techniques to the elimination of these molecules. The secondary objective is to describe and compare the therapeutic therapies adopted in the Intensive Care Units participating in the project.

For each molecule, the study will involve 300 patients admitted to Intensive Care Units. For each patient five blood samples will be collected on average, in order to measure drug plasma concentrations. Patient clinical conditions will be collected through an electronic clinical record. Finally, on the basis of those data, pharmacokinetic models will be developed to describe the evolution in time of drug plasma concentrations.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing antibiotic therapy with amikacin, linezolid, meropenem, piperacillin/tazobactam, or vancomycin.
* patients whose antibiotic therapy started during the stay in ICU or less than 24h before admission to ICU.
* patients with anticipated length of stay in ICU of at least 24h.
* patients with already-placed catheter

Exclusion Criteria:

* patients undergoing antibiotic prophylaxis
* lack of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to Intensive Care Unit (ICU)
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2020-06-26 (Actual); Study Completion 2020-06-26 (Actual)

PRIMARY OUTCOMES:
Drug plasma concentration (time-dependent antibiotics) | 30 min after first dose; 1 day after first dose; 2 day after first dose; 2 measures between the 3rd and the 8th day of treatment
Drug plasma concentration (concentration-dependent antibiotics) | 30 min after first dose; immediately before second dose; peak and trough of the same dose in the 2nd day of therapy; peak and trough of the same dose between the 3rd and the 5th day of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Finazzi, PhD, Principal Investigator — Mario Negri Institute for Pharmacological Research; Elena Garbero, M.Sci, Principal Investigator — Mario Negri Institute for Pharmacological Research
Locations (11):
- Italy (11):
  - Ospedale Maurizio Bufalini, UO Anestesia Terapia Intensiva, Cesena, Emilia-Romagna
  - Ospedale S. Giovanni di Dio ASL 10, Servizio Anestesia e Rianimazione, Florence, FI
  - Ospedale San Giovanni di Dio, Orbetello, Grosseto
  - Presidio Ospedaliero "San Leopoldo Mandic", Merate, Lecco
  - Ospedale A. Manzoni, U.O. Anestesia e Rianimazione 1, Lecco, Lombardy
  - Ospedale San Giovanni Bosco, Servizio Anestesia e Rianimazione B-DEA, Turin, Piedmont
  - Fondazione IRCCS Policlinico San Matteo, Pavia, PV
  - Ospedale del Mugello, Borgo San Lorenzo, Tuscany
  - Ospedale Santa Maria Nuova, Anestesia e Rianimazione, Florence, Tuscany
  - Ospedale Maggiore, C.A. Pizzardi, Bologna
  - Ospedale Misericordia, Grosseto